CLINICAL TRIAL: NCT04676789
Title: Anti-PD-1 Antibody and Pegaspargase Combined With Radiotherapy As First-Line Treatment in Early-Stage Extranodal Natural Killer/T Cell Lymphoma, Nasal Type (ENKTL)
Brief Title: Anti-PD-1 Antibody and Pegaspargase Combined With Radiotherapy in Early-Stage ENKTL
Acronym: SPENT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wanghua, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-ENKTL-002
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
Keywords: sintilimab; Pegaspargase; Definitive intensity-modulated radiotherapy (IMRT)
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — pegaspargase; spartalizumab; sintilimab

STUDY DESIGN:
Intervention Model Description: treatment with sintilimab and pegaspargase combined with intensity-modulated radiotherapy (IMRT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/treatment (Experimental): Patients will receive sintilimab,200mg,ivdrip,day1; pegaspargase,2,500 unit/m2 deep intramuscular injection at three different sites,day 1, every 3 weeks for 4 cycles before radiation.Definitive intensity-modulated radiotherapy (IMRT) will be given. Concurrent sintilimab of 200mg and pegaspargase,2,500 unit/m2 will be administered every 3 weeks for 2 cycles during IMRT for patients who do not achieve complete remission to previous induction therapy. After radiotherapy or CCRT, patients achieving CR with positive plasma EBV-DNA or partial response will continue with sintilimab maintenance up to 2 years.
  Interventions: Drug: Pegaspargase; Drug: Anti-PD-1 monoclonal antibody; Radiation: Definitive intensity-modulated radiotherapy (IMRT)

INTERVENTIONS:
Drug: Pegaspargase — Pegaspargase 2500IU/m2 administered by intramuscular injection on Day 1
  Other Names: P-ASP
Drug: Anti-PD-1 monoclonal antibody — Anti-PD-1 antibody 200mg administered intravenously (IV) on Day 1
  Other Names: sintilimab
Radiation: Definitive intensity-modulated radiotherapy (IMRT) — Definitive intensity-modulated radiotherapy (IMRT) of 50 Gy will be given in 25 days
  Other Names: IMRT

SUMMARY:
Aim of the trial is to evaluate the safety and efficacy of sintilimab and pegaspargase in combination with pegaspargase for the initial treatment of previously untreated patients with limited stage NK/T cell lymphoma.All eligible patients will be treated with sintilimab combined with pegaspargase administered every 3 weeks for 4 cycles followed by standard radiotherapy with or without concurrent sintilimab and pegaspargase administered every 3 weeks. After radiotherapy, patients with complete remission with positive plasma EBV-DNA or partial response will continue with sintilimab maintenance up to 2 years.

DETAILED DESCRIPTION:
This is a multicentre, open-label, single-arm, phase II clinical study to evaluate the safety and efficacy of sintilimab and pegaspargase in combination with pegaspargase for the initial treatment of previously untreated patients with limited stage NK/T cell lymphoma.All eligible patients will be firstly treated with sintilimab combined with pegaspargase administered every 3 weeks for 4 cycles. If the patient achieves complete remission（CR）, standard radiotherapy will be performed, otherwise, they will receive concurrent chemoradiotherapy（CCRT）(radiation 50 Gy and two cycles of sintilimab and pegaspargase every 3 weeks). After radiotherapy or CCRT, patients achieving CR with positive plasma EBV-DNA or partial response will continue with sintilimab maintenance up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ENKTL
* age:18-80years
* Ann Arbor stage IE,or stage IIE
* at lease one measurable lesion
* receive no chemotherapy or radiotherapy before
* Eastern CooperativeOncology Group performance status of 0 to 2.
* Adequate hematologic function (eg, white blood cell ≥ 3×10e9/l,neutrophils count ≥1.5×10e9/L, and platelet count≥ 100×10e9/L),renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria
* non-nasal type disease
* systematic central nervous system involvement
* previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | Baseline up to data cut-off (up to approximately 4 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
complete remission (CR) rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria and 2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy.
overall response rate (ORR) | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria and 2016 Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy.
overall survival (OS) | Baseline up to data cut-off (up to approximately 4 years)
  Overall survival in the overall study population was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event.
Duration of response | Baseline up to data cut-off (up to approximately 4 years)
  Time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with PET-CT.
EBV-DNA load change | At the end of Cycle 6 (each cycle is 21 days)
  EBV-DNA load at each cycle for comparison
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Baseline up to data cut-off (up to approximately 4 years)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, MD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Please Select, China